CLINICAL TRIAL: NCT00701571
Title: Video/Audio Distraction Analgesia for Simulated Oncology Procedure Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Seattle Cancer and Aging Program (Unknown)
Responsible Party: Principal Investigator, Chris Hoffer, Research Coordinator, University of Washington
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 26745; 1R21CA107256-01A1 (NIH); P20CA103728-04 (NIH)
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Last update posted 2011-09-13 (Estimated); Status verified 2011-09

CONDITIONS: Pain
Keywords: Virtual Reality; Oncology; Lumbar puncture
MeSH Terms: conditions — Pain; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): 3 cohorts: 18-21 years, 40-60 years, and older than 60 years
  Interventions: Procedure: Virtual Reality distraction

INTERVENTIONS:
Procedure: Virtual Reality distraction — Virtual Reality involves the participant wearing a helmet with sight and sound. the visual provided is a type of immersive video game, the game used is "Snow World". In some cases the participant will be exposed to 3D representation of the game, and in other cases a lower tech version with less immersive qualities.

SUMMARY:
The purpose of this study is to compare the analgesic efficacy of three different types of video/audio distraction in normal volunteers subjected to carefully controlled and non-injurious thermal pain delivered to the skin of the lower back, simulating discomfort of a lumbar puncture. Two of the distraction techniques include immersive virtual reality (VR). The most efficacious distraction technique will be used in a subsequent clinical study in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* healthy men and women
* 18-21y, 40-60y, or older than 60y

Exclusion Criteria:

* a predisposition to motion sickness
* unusual sensitivity or lack of sensitivity to pain
* chronic pain
* peripheral neuropathy
* sensitive skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2005-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To compare positional techniques and differing types of VR presentation (immersive vs. low tech). We will also compare age cohorts (18-21, 40-60, and older than 60 years). | upon completion of data collection

CONTACTS AND LOCATIONS:
Overall Officials: Samuel R Sharar, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States